CLINICAL TRIAL: NCT00482313
Title: A Single Centre, Randomised, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate Efficacy of PR OROS Methylphenidate Followed by Open-Label Extension, in Swedish Male Prison Inmates With ADHD
Brief Title: Efficacy and Effectiveness of Methylphenidate in Swedish Male Prison Inmates With Attention-deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Psychiatry Karolinska (Other)
Collaborators: Ministry of Health and Social Affairs, Sweden (Other Government); Region Stockholm (Other Government)
Responsible Party: Nils Lindefors, MD, PhD, Karolinska Institutet, Psychiatry Southwest, Karolinska University Hospital at Huddinge, Stockholm, Sweden
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCT-nr 2006-002553-80
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Last update posted 2010-05-10 (Estimated); Status verified 2009-08

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; ADHD; Prison; Treatment; Randomized; Double-Blind; Placebo Control; Parallel Assignment; Efficacy Study
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylphenidate (Experimental): PR OROS Methylphenidate given orally once daily for 5 weeks. The dosage was as follows: 36 mg per day from day 1-3, 54 mg per day from day 4-7 and 72 mg per day from day 8 until end of 5th week.
  Interventions: Drug: PR OROS Methylphenidate
- Sugar pill (Placebo Comparator): Placebo given orally once daily for 5 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PR OROS Methylphenidate — PR OROS Methylphenidate given orally once daily for 5 weeks. The dosage was as follows: 36 mg per day from day 1-3, 54 mg per day from day 4-7 and 72 mg per day from day 8 until end of 5th week.
  Other Names: Concerta
  Arms: Methylphenidate
Drug: Placebo — Sugar pill
  Arms: Sugar pill

SUMMARY:
The purpose of this study is to evaluate the efficacy and effectiveness of methylphenidate in treatment of ADHD in Swedish adult male prison inmates diagnosed with ADHD.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy of Prolonged Release (PR) OROS methylphenidate in fixed dosage as compared to placebo, and the effectiveness of flexible dosage Prolonged Release (PR) OROS methylphenidate in Swedish adult male prison inmates with attention-deficit hyperactivity disorder (ADHD). An initial randomised, double-blind, placebo-controlled parallel group trial for 5 weeks is followed by an open-label extension for maximum 47 weeks, comprising altogether 52 weeks of treatment. A follow-up is carried out 12 and 36 months post-study, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Male, 18-65 years, imprisoned at Norrtalje Prison
* WURS-score of 36 or more and fulfilling at least 4 out of 6 criteria on ASRS Screener in an initial screening preceding the trial
* Can read and understand Swedish well enough to participate in the evaluation preceding the trial
* Diagnosis of ADHD according to the Diagnostic and Statistical Manual of Mental Diseases, Fourth Edition, (DSM-IV) and confirmed by the neuropsychiatric assessment including structured diagnostic interviews and neuropsychological measurements.
* At least 14 months left to conditional release.
* Informed Consent Form to participate in the study signed by the subject.
* Subject agrees to take only the supplied study drug as treatment for ADHD during the study
* Subject is able to comply with the study visit schedule and willing and able to complete the protocol-specified assessments.
* Healthy on the basis of a physical examination and the results of blood biochemistry tests. If the results of the biochemistry tests are not within the normal reference ranges, the subject may be included if the investigator considers the deviations are not clinically relevant.

Exclusion Criteria:

* Known to be a non-responder to methylphenidate.
* Known allergy or hypersensitivity to methylphenidate.
* Any clinically unstable psychiatric condition including, but not limited to, acute mood disorder, bipolar disorder, acute OCD.
* A diagnosis of substance use disorder (abuse/dependence) according to DSM-IV criteria within 3 months prior to screening evaluation for the study.
* Known mental retardation.
* Subjects with history of epileptic seizures, glaucoma, uncontrolled hypertension, angina pectoris, cardiac arrhythmias or structural heart abnormalities.
* Use of monoamine oxidase inhibitors, fluoxetine, venlafaxine, reboxetine, duloxetine.
* Use of alpha-2-receptor agonists, neuroleptics, theophylline, coumarin anticoagulants or anticonvulsants.
* Liver or renal insufficiency. Subjects with hepatitis C without liver insufficiency don´t have to be excluded as long as liver enzymes are followed through the study.
* Subjects who are suicidal.
* Lactose intolerance.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-05; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Efficacy of PR OROS methylphenidate on ADHD-symptoms in adult male prison inmates with ADHD, as measured by changes from baseline until endpoint in the observer-rated CAARS. | Changes from baseline until endpoint at week 5
  ADHD-symptoms as measured by changes in the observer-rated CAARS from baseline until endpoint at week 5.

SECONDARY OUTCOMES:
Long-term effectiveness of PR OROS methylphenidate as measured by changes from baseline until endpoint in ADHD-symptoms, global functioning, neuropsychological functioning, and quality of life in adult male prison inmates with ADHD. | From baseline until endpoint at week 52
  ADHD-symptoms as measured by changes in the observer-rated CAARS, and by the self-reported ASRS until endpoint at week 52.
  Global functioning as measured by changes in CGI-S and GAF until endpoint at week 52.
  Neuropsychological functioning, as measured by changes in the Conners CPT II, the QbTestPlus, Digit Span and Span Board from baseline until endpoint at week 52.
  Quality of Life as measured by changes in the Quality of Life Inventory from baseline until endpoint at week 52.
Efficacy of PR OROS methylphenidate on ADHD-symptoms and global functioning in adult male prison inmates with ADHD, as measured by changes from baseline until endpoint in self-reported ASRS, CGI-S and GAF | From baseline until endpoint at week 5
Safety parameters, as measured by changes in pulse, blood pressure, weight and blood chemistry, from baseline until endpoint. | From baseline until endpoint at week 52
  Blood chemistry included counting of red blood cells, white blood cells, blood platelets, and liver enzymes (ALAT, ASAT).
Safety parameters as collection of reported adverse events from baseline until endpoint | From baseline until endpoint at week 52

CONTACTS AND LOCATIONS:
Overall Officials: Nils Lindefors, MD, PhD, Principal Investigator — Karolinska Institutet, Psychiatry Southwest, Karolinska University Hospital at Huddinge, Stockholm, e-mail: nils.lindefors@sll.se
Locations (1):
- Stockholm County Council, Psychiatry Southwest Karolinska, Huddinge, Stockholm County, Sweden

REFERENCES:
- [Derived] Ginsberg Y, Langstrom N, Larsson H, Lindefors N. Long-Term Treatment Outcome in Adult Male Prisoners With Attention-Deficit/Hyperactivity Disorder: Three-Year Naturalistic Follow-Up of a 52-Week Methylphenidate Trial. J Clin Psychopharmacol. 2015 Oct;35(5):535-43. doi: 10.1097/JCP.0000000000000395. PMID 26284932
- [Derived] Ginsberg Y, Lindefors N. Methylphenidate treatment of adult male prison inmates with attention-deficit hyperactivity disorder: randomised double-blind placebo-controlled trial with open-label extension. Br J Psychiatry. 2012 Jan;200(1):68-73. doi: 10.1192/bjp.bp.111.092940. Epub 2011 Nov 10. PMID 22075648